CLINICAL TRIAL: NCT05735314
Title: A New Combination of Evidence-Based Interventions to Improve Primary Care Diagnostic Safety and Efficiency: a Stepped Wedge Cluster Randomized Control Trial (RCT)
Brief Title: A New Combination of Evidence-Based Interventions to Improve Primary Care Diagnostic Safety and Efficiency
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Eric Thomas, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: HSC-MS-22-0815
Record Dates: First submitted 2023-02-07; First posted 2023-02-21 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Anemia; Decreased Glomerular Filtration Rate
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Intervention Model Description: This is a stepped wedge cluster-randomized trial. There will be 4 clusters, with 3-4 clinics per cluster. In a stepped wedge fashion, the 4 clusters will receive the control followed by the study intervention--that is, in the first step the first cluster will receive the intervention after 6 months of control, in the second step the second cluster will receive intervention after 12 months of control, in the third step the third cluster will receive the intervention after 18 months of control, and in the fourth step the fourth cluster will receive the intervention after 24 months of control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental: Step 1 (3 clinics) - 24 months of intervention (Experimental)
  Interventions: Other: Enhanced diagnostic team implementing three evidence-based interventions; Other: Usual care
- Experimental: Step 2 (3 clinics) - 1 month of control followed by 18 months of intervention (Experimental)
  Interventions: Other: Enhanced diagnostic team implementing three evidence-based interventions; Other: Usual care
- Experimental: Step 3 (3 clinics) - 2 months control followed by 12 months of intervention (Experimental)
  Interventions: Other: Enhanced diagnostic team implementing three evidence-based interventions; Other: Usual care
- Experimental: Step 4 (4 clinics) - 2 months control followed by 12 months of intervention (Experimental)
  Interventions: Other: Enhanced diagnostic team implementing three evidence-based interventions; Other: Usual care

INTERVENTIONS:
Other: Enhanced diagnostic team implementing three evidence-based interventions — we designed an enhanced team process entailing: 1) using automated abnormal test result detection and tracking; 2) expanding the primary care team to include CPs to guide the evaluation of anemia to identify underlying causes; and 3) using NNs to engage patients in the healthcare team and diagnostic process and increase patient activation.
Other: Usual care — Usual care involves primary care physicians ordering additional tests and referrals to evaluate patients with new anemia and decreased glomerular filtration rate (GFR) .
  Other Names: Control

SUMMARY:
The purpose of this study is to measure the evidence-based intervention's (EBIs) impact on patient safety and efficiency, to assess the EBIs implementation by measuring acceptability, appropriateness, cost, fidelity, penetration, and sustainability and to identify the facilitators and barriers that influence the degree of implementation of these EBIs.

ELIGIBILITY:
Primary care providers' inclusion criteria:

* physicians, physicians assistants and advanced practice registered nurses in the 13 clinic locations of UTP are eligible if they care for patients at the time patient enrollment at their clinic begins
* agree to participate.

Patients' inclusion criteria are:

* hemoglobin result < 10.8 for females and < 12.5 for males with normal white cell count and platelet count (the prior hemoglobin results must have been in normal range, with a look-back period of two years)
* an eGFR value < 60 (the prior eGFR results must have been in normal range, with a look-back range of two years)
* the matching creatinine results must also be in normal range
* not pregnant
* speak English or Spanish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2026-07-16 (Estimated); Study Completion 2026-07-16 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects who have correct diagnosis of cause of low hemoglobin | within 6 months from baseline
  Percentage of subjects who have correct diagnosis of cause of low hemoglobin
Percentage of subjects who have correct diagnosis of cause of low glomerular filtration | within 6 months from baseline
  Percentage of subjects who have correct diagnosis of cause of low glomerular filtration

SECONDARY OUTCOMES:
Time until diagnosis | initial abnormal test result to the day the diagnosis was communicated to the patient (about 1-6 months)
  Time until diagnosis is defined as number of days from the initial abnormal test result to the day the diagnosis was communicated to the patient.
Percentage of tests appropriately utilized | within 6 months from baseline
  Percentage of tests appropriately utilized will be calculated as the number of appropriate tests ordered to evaluate the abnormal test divided by the total number of tests ordered to evaluate the abnormal test, multiplied by 100.
Cost of treatment | from baseline to 6 months
  Costs will be assessed from the health care system perspective and will include the costs of all diagnostic tests and referral consultations to evaluate the abnormal tests, emergency department (ED) visits or admissions for care for the underlying diseases causing test abnormalities, and the personnel time to provide the EBIs during the 6-month work up period.
Number of primary care physicians (PCPs) who find the intervention as acceptable assessed by survey of PCPs | 12 weeks after PCP's patient enrolled
  Number of primary care physicians (PCPs) who find the intervention as acceptable
Number of PCPs who find the intervention appropriate as assessed by survey of PCPs | 12 weeks after PCP's patient enrolled
  Number of PCPs who find the intervention appropriate as assessed by survey of PCPs
Number of PCPs who find the intervention feasible as assessed by survey of PCPs | 12 weeks after PCP's patient enrolled
  Number of PCPs who find the intervention feasible as assessed by survey of PCPs
Fidelity as assessed by the percentage of participants who moved through each step of the diagnostic process needed for their diagnosis | 6 months
  Fidelity as assessed by the percentage of participants who moved through each step of the diagnostic process needed for their diagnosis
Penetration as assessed by the percentage of participants with abnormal tests who receive the intervention | 6 months
  Penetration as assessed by the percentage of participants with abnormal tests who receive
Sustainability as assessed by number of clinics that continued the intervention | 2.5 years
Patient activation as assessed by the short form of the Patient Activation Measure (PAM) | between 1 to 6 months
  This 13-item survey uses a 5-point Likert scale to measure 4 domains related to patient activation. Total score ranges from 1 to 65, with a higher score indicating greater activation.
Number of clinics with more facilitators than barriers | 6 months
  Number of clinics with more facilitators than barriers

CONTACTS AND LOCATIONS:
Overall Officials: Eric Thomas, MD,MPH, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Novikov Z, Mehra N, Li X, Wells R, Ottosen M, Hwang K, Avritscher EBC, Green C, Lee KH, Oguin X, Janecka M, Espinoza M, Adebowale B, Araya A, Wahed A, Thomas E. Evidence-based team intervention to reduce diagnostic errors in anaemia and CKD diagnoses in primary care: protocol for a stepped-wedge cluster RCT. BMJ Open. 2026 Feb 5;16(2):e112391. doi: 10.1136/bmjopen-2025-112391. PMID 41644166